CLINICAL TRIAL: NCT04820777
Title: Effects Of Perturbation Based Balance Training in Reactive Balance Control Among Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2049 Hira Irfan
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Stroke; Perturbation based training; Fall; Berg balance scale; Performance oriented mobility assessment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perturbation based training (Experimental): External perturbations occur by forces outside the patient' control (e.g., a push or pull from the physiotherapist). Internal perturbations caused when the patient is unable to control the centre of mass and the base of support relationship during voluntary movement; 'agility' tasks, such as kicking a soccer ball,
  Interventions: Other: perturbation training
- Conventional' balance training (Active Comparator): Starting from a situated position, expand your left leg until it's corresponding to the floor. Try not to bolt your knee. At that point, gradually bring your foot down to the floor.
  Rehash with your correct leg, exchanging to and fro between legs for a sum of 20 repitions (10 on every leg).
  Situated Marching Starting with a situated position, lift your effected leg towards your chest, making an honest effort to keep up controlled development.
  Interventions: Other: Conventional' balance training

INTERVENTIONS:
Other: perturbation training — external or internal postural perturbations. External perturbations occur by forces outside the patient' control (e.g., a push or pull from the physiotherapist). Internal perturbations caused when the patient is unable to control the centre of mass and the base of support relationship during voluntary movement; 'agility' tasks, such as kicking a soccer ball,
  Arms: perturbation based training
Other: Conventional' balance training — Starting from a situated position, expand your left leg until it's corresponding to the floor. Try not to bolt your knee. At that point, gradually bring your foot down to the floor. Rehash with your correct leg, exchanging to and fro between legs for a s
  Arms: Conventional' balance training

SUMMARY:
Chronic stroke patients often have impaired balance on reactive balance control. Task specific exercises are important part of the fall intervention in daily activities of life should be incorporated during the rehabilitative services Objective: Effects of perturbation based balance training in reactive balance control in chronic stroke patients.

DETAILED DESCRIPTION:
RCT (Randomized Control Trail) study was conducted. Stroke patients who have impaired balance and reactive control were determined on inclusion & exclusion criteria. Stroke patients with impaired balance control were arbitrarily allocated into two groups with one control and one interventional group ages ranged from 45 to 50 years. The sample size was 20 patients. Group 1 (control group) received tradional balance training and Group 2 (interventional group) received perturbation based training for balance control. The interval of treatment was 6 weeks. Data is collected from Azra Naheed Medical college (Ch Muhammad Akram teaching & research hospital) Lahore and Physiotherapy department of Social security hospital manga mandi Lahore. Tinetti performance oriented mobility assessment (POMA),Time up and go (TUG) and Activity specific balance confidence (ABC) was used to evaluate the pre and post values of balance control.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who was not obese and BMI was <28
* Individuals at chronic stroke level (>6 months post stroke).
* The patients who can walk with or without a gait aid (but without assistance of another

Exclusion Criteria:

* • Different neurological diseases and problems that can impaired balance control (e.g. Parkinson's disease); upper or the lower body parts amputation; cognitive, language, or social impairments which can affect the following of instructions.

  * Patients who were attending any perturbation based training
  * Patients who were visually impaired, having orthostatic hypotension or dizziness

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Tinetti performance oriented mobility assessment | 2 months
  POMA for gait and balance for stroke patients
Time up and go (TUG) | 2 months
  screening test that is a sensitive and specific measure of probability for falls among older adults[
Activity specific balance confidence (ABC) | 2 months
  the Activities-specific Balance Confidence Scale (ABC Scale) is a structured questionnaire that measures an individual's confidence in performing activities without losing balance

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Duijnhoven HJ, Heeren A, Peters MA, Veerbeek JM, Kwakkel G, Geurts AC, Weerdesteyn V. Effects of Exercise Therapy on Balance Capacity in Chronic Stroke: Systematic Review and Meta-Analysis. Stroke. 2016 Oct;47(10):2603-10. doi: 10.1161/STROKEAHA.116.013839. Epub 2016 Sep 15. PMID 27633021
- [Background] In T, Lee K, Song C. Virtual Reality Reflection Therapy Improves Balance and Gait in Patients with Chronic Stroke: Randomized Controlled Trials. Med Sci Monit. 2016 Oct 28;22:4046-4053. doi: 10.12659/msm.898157. PMID 27791207
- [Background] Lund C, Dalgas U, Gronborg TK, Andersen H, Severinsen K, Riemenschneider M, Overgaard K. Balance and walking performance are improved after resistance and aerobic training in persons with chronic stroke. Disabil Rehabil. 2018 Oct;40(20):2408-2415. doi: 10.1080/09638288.2017.1336646. Epub 2017 Jun 9. PMID 28597708
- [Background] Vahlberg B, Cederholm T, Lindmark B, Zetterberg L, Hellstrom K. Short-term and long-term effects of a progressive resistance and balance exercise program in individuals with chronic stroke: a randomized controlled trial. Disabil Rehabil. 2017 Aug;39(16):1615-1622. doi: 10.1080/09638288.2016.1206631. Epub 2016 Jul 14. PMID 27415645
- [Background] Lee D, Lee G. Effect of afferent electrical stimulation with mirror therapy on motor function, balance, and gait in chronic stroke survivors: a randomized controlled trial. Eur J Phys Rehabil Med. 2019 Aug;55(4):442-449. doi: 10.23736/S1973-9087.19.05334-6. Epub 2019 Mar 22. PMID 30916531
- [Background] Alghadir AH, Al-Eisa ES, Anwer S, Sarkar B. Reliability, validity, and responsiveness of three scales for measuring balance in patients with chronic stroke. BMC Neurol. 2018 Sep 13;18(1):141. doi: 10.1186/s12883-018-1146-9. PMID 30213258
- [Background] Tally Z, Boetefuer L, Kauk C, Perez G, Schrand L, Hoder J. The efficacy of treadmill training on balance dysfunction in individuals with chronic stroke: a systematic review. Top Stroke Rehabil. 2017 Oct;24(7):539-546. doi: 10.1080/10749357.2017.1345445. Epub 2017 Jul 7. PMID 28687056
- [Background] Liu TW, Ng GYF, Ng SSM. Effectiveness of a combination of cognitive behavioral therapy and task-oriented balance training in reducing the fear of falling in patients with chronic stroke: study protocol for a randomized controlled trial. Trials. 2018 Mar 7;19(1):168. doi: 10.1186/s13063-018-2549-z. PMID 29514677
- [Background] Sharma V, Kaur J. Effect of core strengthening with pelvic proprioceptive neuromuscular facilitation on trunk, balance, gait, and function in chronic stroke. J Exerc Rehabil. 2017 Apr 30;13(2):200-205. doi: 10.12965/jer.1734892.446. eCollection 2017 Apr. PMID 28503533
- [Background] Schinkel-Ivy A, Huntley AH, Aqui A, Mansfield A. Does Perturbation-Based Balance Training Improve Control of Reactive Stepping in Individuals with Chronic Stroke? J Stroke Cerebrovasc Dis. 2019 Apr;28(4):935-943. doi: 10.1016/j.jstrokecerebrovasdis.2018.12.011. Epub 2019 Jan 7. PMID 30630753